CLINICAL TRIAL: NCT06792422
Title: Additive Benefits of Semaglutide for Open-AngLe Glaucoma - an Opportunity for Neuroprotection
Brief Title: A Study Investigating Oral Semaglutide in People with Open-Angle Glaucoma
Acronym: ABSALON
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Miriam Kolko, Professor in Translational Eye Research, Chief Physician., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 97669; NNF22OC0079544 (Other Grant/Funding Number: The Novo Nordisk Foundation); 2024-518510-87-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-18; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-11

CONDITIONS: Primary Open Angle Glaucoma (POAG); Open-Angle Glaucoma; Glaucoma
Keywords: Glaucoma; Semaglutide; Rybelsus; Primary Open Angle Glaucoma; GLP-1RA; Photopic Negative Response; GLP-1
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Semaglutide (Experimental): Participants are given oral semaglutide once daily.
  Interventions: Drug: Oral semaglutide
- Placebo (Placebo Comparator): Participants are given oral placebo once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral semaglutide — Participants will receive oral semaglutide once daily.
  1. Starting dose 3 mg/day for one month (day 1-28)
  2. Intermediate dose 7 mg/day for one month (day 29-56)
  3. Maintenance dose 14 mg/day (day 57-182)
  Arms: Oral Semaglutide
Drug: Placebo — Participants will receive an oral placebo once daily.
  1. Placebo tablets received on visit 1 (baseline) for one month (day 1-28)
  2. Placebo tablets received on visit 2 (month 1) for one month (day 29-56)
  3. Placebo tablets received on visit 3 (month 2) for four months (day 57-182)
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to investigate whether oral semaglutide can be used to treat open-angle glaucoma. The main question it aims to answer is: Does oral semaglutide safely improve inner retinal function in patients with open-angle glaucoma as measured by the photopic negative response of the electroretinogram.

Researchers will compare oral semaglutide to a placebo (a look-alike substance that contains no drug).

Participants will:

* Take semaglutide or a placebo every day for 6 months.
* Visit the clinic 5 times in total for tests and interviews: At baseline (the first day they are included in the study), after 1 month, after 2 months, after 3 months, and after 6 months (the last day they are included in the study).

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and speak Danish
* 45 years or older at the time of inclusion
* Visual acuity equal to or above 0.5 in the study eye
* Diagnosis of POAG with MD ≤ 16 dB with repeatable and reliable (false positive less than 15 %) VF loss measured by standard automated perimetry on at least one eye
* Receiving IOP-lowering glaucoma treatment
* Nerve fiber layer defects identified by OCT

Exclusion Criteria:

* Diabetes or renal impairment
* Medical history of significant eye disease (including ocular trauma) other than glaucoma
* Ocular inflammation/infection within three months from inclusion
* Intraocular surgery 3 months before inclusion
* Smoker at the time of inclusion
* Pregnant or breast-feeding
* Females of childbearing potential who are not using adequate contraceptive, which includes the following: Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal, progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, or implantable; Intrauterine device (IUD); Intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomised partner; Sexual abstinence
* Subjects allergic to drug ingredients administered during the trial
* Subjects with untreated severe systemic disease or malignancies
* Previous history of pancreatitis
* BMI < 18.5
* Subjects receiving treatment with: Dipeptidyl peptidase-4 inhibitors; Other GLP-1RAs; Insulin; Insulin analogues; Sulfonylurea; Systemic corticosteroids; Immunosuppressants

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 126 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Photopic negative response of the electroretinogram after 6 months | From baseline to month 6.
  Change in the inner retinal function assessed by mean change in the photopic negative response of the electroretinogram.

SECONDARY OUTCOMES:
Photopic negative response of the electroretinogram after 3 months | From baseline to month 3.
  Change in the inner retinal function assessed by mean change in the photopic negative response of the electroretinogram.
Pelli-Robson chart contrast sensitivity test | From baseline to month 6.
  Functional glaucoma progression assessed using the Pelli-Robson chart contrast sensitivity test.
Health-related quality of life (HRQoL) | From baseline to month 6.
  Health-related quality of life (HRQoL) assessed with the European Quality of life - 5 Dimensions - 3 Levels (EQ-5D-3L) questionnaire, a standardized validated questionnaire administered in Danish. The EQ-5D-3L questionnaire comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Health-related quality of life (HRQoL) | From baseline to month 6.
  Health-related quality of life (HRQoL) assessed with the 25-item National Eye Institute Visual Function Questionnaire (NEI VFQ-25), a standardized validated questionnaire administered in Danish. The scoring system for the NEI VFQ-25 generates 12 subscale scores and an overall composite score. A higher score indicates a higher level of functioning.
Number of treatment-related adverse events as assessed by CTCAE v5.0 | From baseline to month 6.
  Safety and tolerance of oral semaglutide treatment in patients with glaucoma assessed by the incidence of treatment-emergent adverse events (TEAEs) by CTCAE v5.0.

OTHER OUTCOMES:
Optical coherence tomography (OCT), ring scan | From baseline to month 6.
  Structural glaucoma progression assessed by the OCT ring scan, which measures the retinal nerve fibre layer thickness.
Optical coherence tomography (OCT), macular scan | From baseline to month 6.
  Structural glaucoma progression assessed by the OCT macular scan which measures the volume of retinal ganglion cells.
Standard automated perimetry | From baseline to month 6.
  Visual field loss will be evaluated using standard automated perimetry. Progression will be measured by changes in mean deviation (MD).
Multi-omics | From baseline to month 6.
  Changes in the cytokine proteome will be assessed by changes in concentrations of glaucoma-associated cytokines as related to inflammation. Changes in the metabolome and lipidome will be assessed by changes in plasma metabolomics and lipidomics.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Rigshospitalet, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No